CLINICAL TRIAL: NCT05403749
Title: A Multi-center, Randomized, Double-masked, Active-controlled Study to Evaluate the Longer Interval of Intravitreal (IVT) Injection of IBI302 in Subjects With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: A Study of Longer Interval of IVT IBI302 in Subjects With nAMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI302A202
Record Dates: First submitted 2022-05-20; First posted 2022-06-03 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI302 dose 2 group (Experimental): Drug: Aflibercept 8mg/eye;Intraocular injection
  Interventions: Biological: dose 2 IBI302
- Aflibercept (Active Comparator): Drug: Aflibercept 2mg/eye;Intraocular injection
  Interventions: Drug: Aflibercept
- IBI302 dose 1 group (Experimental): Drug: Aflibercept 6.4mg/eye;Intraocular injection
  Interventions: Biological: dose 1 IBI302

INTERVENTIONS:
Biological: dose 1 IBI302 — After 4 loading monthly intravitreal injections of dose 1 IBI302，the following IBI302 IVT is given as descript in protocol.
  Arms: IBI302 dose 1 group
Drug: Aflibercept — Three consecutive monthly intravitreal injections of 2.0mg Aflibercept followed by injection every other month
  Arms: Aflibercept
Biological: dose 2 IBI302 — After 4 loading monthly intravitreal injections of dose 2 IBI302，the following IBI302 IVT is given as descript in protocol
  Arms: IBI302 dose 2 group

SUMMARY:
The study is designed for multi-center, randomized, double-masked, active-controlled study to evaluate the longer interval of intravitreal injection of IBI302 in subjects with neovascular age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign informed consent from and comply with visit and study procedures per protocol.
2. Male or female patients≥50 yrs. of age.
3. Active subfoveal or parafoveal CNV secondary to neovascular AMD on FFA or OCT.
4. The CNV area≥50% lesion area on FFA in the study eye at screening visit.
5. BCVA score of 24-78 letters using ETDRS charts in the study eye at the baseline.

Exclusion Criteria:

1. Concomitant diseases that may cause subjects fail to respond to the treatment or confuse the interpretation of the study results.
2. Subretinal hemorrhage>50% total lesion area and/or involvement in the macular foveal, fibrosis or atrophy area>50% total lesion area and/or involved of macular fovea;
3. Presence of uncontrolled glaucoma in the study eye(defined as IOP≥25mmHg, or judged by the investigators at the screening or baseline visit)
4. Presence of active intraocular or periocular inflammation or infection;
5. Prior any treatment of following in the study eye:

   * Anti-VEGF(Vascular Endothelial Growth Factor) therapy or anti-complement therapy within 3 months prior to screening;
   * Laser photocoagulation within 3 months prior to screening;
   * Photodynamic therapy or vitreoretinal surgery;
   * Intraocular glucocorticoid injection within 6 months prior to enrollment;
6. Presence of any systemic disease: including but not limited tractive infections (such as active viral hepatitis); unstable angina; cerebrovascular accident or transient cerebral ischemia (within 6 months prior to selection); myocardial infarction (within 6 months prior to selection); serious arrhythmia requiring medical treatment; liver, kidney or metabolic diseases; or malignant tumor;
7. History of severe hypersensitivity/allergy to active ingredients or any excipients of the study drug, or fluorescein and povidone iodine;
8. Pregnant or lactating women or women preparing to become pregnant or breastfeeding during the study period;
9. Participated in any clinical study of any other drug within three months prior to enrollment, or attempted to participate in other drug trials during the study;
10. Other conditions unsuitable for enrollment judged by investigators

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Change of BCVA from baseline | Baseline to week 40
  Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.

SECONDARY OUTCOMES:
Percentage of Participants Loss >0,≥5,10，15 Letters From the Baseline BCVA in the Study Eye Over Time | Baseline to week 52
  Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a loss in BCVA letter score from baseline indicates a decline in visual acuity.
Change of Central Subfield Thickness in the Study Eye from baseline | Baseline to week 52
  Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane using optical coherence tomography (OCT), as assessed by the central reading center.
Change of Total Area of Choroidal Neovascularization (CNV) Lesion/Total Area of Choroidal Neovascularization Leakage in the Study Eye from Baseline | From Baseline to week 52
  The total area of the choroidal neovascularization lesion/Total Area of Choroidal Neovascularization Leakage in the study eye was evaluated by a central reading center using fundus fluorescein angiography (FFA).
Percentage of Participants in different dosage of IBI302 Arm on Once Every 8-Weeks, 12-Weeks,Treatment Intervals | At Week 20,40,52
Safety Summary of the Overall Number of Participants With at Least One Adverse Event by Event Type, in All Participants | From Baseline to week 52
  This safety summary reports the number and percentage of participants who experienced at least one adverse event (AE) during the study. AEs are categorized as any AEs, ocular AEs occurring in the study eye or fellow eye, systemic AEs, serious AEs, AEs related to treatment with study drug, AEs of special interest. The investigator independently assessed the seriousness and severity for each AE. Severity was graded according to the following grading scale: Mild = Discomfort noticed, but no disruption of normal daily activity; Moderate = Discomfort sufficient to reduce or affect normal daily activity; Severe = Incapacitating with inability to work or to perform normal daily activity.
Percentage of Participants Gaining ≥0,5,10,15 Letters From the Baseline BCVA in the Study Eye Over Time | From Baseline to week 52
  Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Immunogenicity end points | From Baseline to week 52
  Production of anti-drug antibodies in serum.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China